CLINICAL TRIAL: NCT03185637
Title: Paediatric Surgery Across Sub-Saharan Africa: A Multi-Centre Prospective Cohort Study
Brief Title: Children's Surgery in Sub-Saharan Africa
Acronym: PaedSurgAfrica
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Sylvanus Olympio University Teaching Hospital, Lome, Togo. (Unknown); National Hospital of Niamey (Other); Centre Hospitalier Universitaire de la Mère et de l Enfant, Cotonou, Benin. (Unknown); HEAL Africa Hospital, Goma, Democratic Republic of the Congo. (Unknown); Centre Hospitalier Universitaire Pédiatrique Charles de Gaulle (Other); University Hospital De Bouaké, Ivory Coast. (Unknown); Teaching Hospital Treichville, Abidjan, Ivory Coast. (Unknown); Harare Central Hospital, Zimbabwe. (Unknown); University Teaching Hospital, Lusaka, Zambia (Other); Mulago Hospital, Uganda (Other); Tikur Anbessa Specialized Hospital, Addis Ababa, Ethiopia. (Unknown); Mbingo Baptist Hospital, Cameroon. (Unknown); Ministry of Health, Ghana (Other Government); Korle-Bu Teaching Hospital, Accra, Ghana (Other); Edna Adan Maternity Hospital, Hargeisa, Somaliland. (Unknown); Embu Level 5 Hospital, Kenya. (Unknown); Tenwek Hospital (Other); Soba University Hospital (Other); Kamuzu Central Hospital (Other); Queen Elizabeth Central Hospital, Blantyre, Malawi (Unknown); Muhimbili National Hospital, Dar es Salaam, Tanzania. (Unknown); Grey's Hospital (Other); Stranger Hospital, Kwazulu-Natal, South Africa. (Unknown); Tygerberg Hospital, South Africa. (Unknown); Clinton Hospital, Johannesburg (Unknown); Charlotte Maxeke Johannesburg Academic Hospital (Unknown); Chris Hani Baragwanath Academic Hospital (Other); East London Hospital Complex, South Africa. (Unknown); Red Cross War Memorial Childrens Hospital (Other); Delta State University Teaching Hospital Ogharra (Unknown); Bowen University Teaching Hospital, Ogbomoso (Unknown); Ondo State Trauma and Surgical Centre (Unknown); Mnamdi Azikiwe University Teaching Hospital (Unknown); University Of Nigeria Teaching Hospital (Network); University of Port Harcourt Teaching Hospital (Other); University College Hospital, Ibadan (Other); Ahmadu Bello University Teaching Hospital (Other); University of Abuja Teaching Hospital (Other); National Hospital, Abuja (Other Government); University of Calabar Teaching Hospital (Unknown); Federal Medical Centre, Abeokuta (Unknown); Federal Medical Centre, Owo (Industry); Benue State University Teaching Hospital (Other); Olabisi Onabanjo University Teaching Hospital (Unknown); University of Ilorin Teaching Hospital (Other); Federal Medical Centre Lokoja (Unknown); Lagos State University (Other); Obafemi Awolowo University Teaching Hospital (Other); Aminu Kano Teaching Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PSA2016/7
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-06

CONDITIONS: Gastroschisis; Anorectal Malformation; Appendicitis; Intussusception; Inguinal Hernia
Keywords: Outcomes; Mortality; Complications; Neonatal surgery; Paediatric surgery; Childrens surgery; Sub-Saharan Africa; Research Collaboration; Gastroschisis; Anorectal malformation; Appendicitis; Intussuception; Inguinal hernia
MeSH Terms: conditions — Gastroschisis; Anorectal Malformations; Appendicitis; Intussusception; Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Gastroschisis: All patients presenting primarily to the institution with gastroschisis during the data collection period will be included in the study.
  Interventions: Procedure: Various interventions for each of the conditions.
- Anorectal malformation: All patients presenting primarily to the institution with anorectal malformation during the data collection period will be included in the study.
  Interventions: Procedure: Various interventions for each of the conditions.
- Appendicitis: All patients under 16-years of age presenting primarily to the institution with appendicitis during the data collection period will be included in the study.
  Interventions: Procedure: Various interventions for each of the conditions.
- Intussusception: All patients under 16-years of age presenting primarily to the institution with intussusception during the data collection period will be included in the study.
  Interventions: Procedure: Various interventions for each of the conditions.
- Inguinal hernia: All patients under 16-years of age undergoing surgery for an inguinal hernia at the institution during the data collection period will be included in the study.
  Interventions: Procedure: Various interventions for each of the conditions.

INTERVENTIONS:
Procedure: Various interventions for each of the conditions. — This is an observational study. Patients were not allocated to different interventions.
  Common interventions for each of the conditions, which will be compared during analysis include the following:
  Gastroschisis - primary operative closure, surgical silo, preformed silo. Anorectal malformation - various types of stoma, anoplasty, PSARP, other. Appendicitis - antibiotics, open appendicectomy, laparoscopic appendicectomy. Intussusception - air enema reduction, hydro-enema reduction, laparotomy. Inguinal hernia - open repair, laparoscopic repair.

SUMMARY:
Background: Five billion people worldwide do not have access to safe, affordable surgical care. A significant proportion live in sub-Saharan Africa (SSA), where up to 50% of the population are children. There is limited literature on neonatal and paediatric surgery in SSA and children's surgery does not appear on any of the National Health Strategic Plans for the 47 independent countries across SSA.

Objectives: To form a collaboration of surgeons and allied health professionals involved in children's surgery across SSA and collectively undertake the largest prospective cohort study of paediatric surgery in this region.

Materials and Methods: Data will be collected via REDCap website on all patients with gastroschisis, anorectal malformation, appendicitis, inguinal hernia and intussusception, during a 1-month period of collaborators choice between October 2016 to April 2017, with a 30-day follow up until the end of May 2017. Estimated study population: 1450 patients from 50 institutions. Full ethical approval has been granted by the host centre; local ethical approval will be required at collaborating centres for participation. All collaborators will be co-authors.

Primary outcome will be in-hospital all-cause mortality. Secondary outcomes will include post-intervention complications. Data will be collected on institutional facilities, patient demographics, duration from condition onset to presentation, peri-operative resuscitation, intervention and outcome.

Differences in outcomes between SSA and benchmark data from high-income countries will be calculated using chi-squared analysis. Multi-level multivariate logistic regression analysis will be used to identify interventions and peri-operative factors associated with improved outcomes; p<0.05 will be deemed significant.

Outcome: Results will be used to advocate for enhanced children's surgical services in SSA. We shall identify context-appropriate interventions associated with improved outcome. The collaboration will help to enhance research capacity in the region.

DETAILED DESCRIPTION:
Introduction

Research Collaboratives

PaedSurg Africa aims to recruit surgeons and allied health professionals undertaking neonatal and paediatric surgery (PS) across sub-Saharan Africa (SSA) - an area heavily neglected in global health prioritisation. Such research collaboratives are being increasingly utilised as a highly effective and efficient method of collecting large volume prospective data in a short period of time. A great recruitment incentive will be ethical group co-authorship of published results for all research collaborators.

Global Paediatric Surgery

In 2015, the Lancet Commission on Global Surgery (LCoGS) highlighted that 5 billion people worldwide do not have access to safe, affordable surgical care. The same year, the World Health Assembly (Resolution 68.15) incorporated emergency and essential surgery and anaesthesic care within 'Universal Health Coverage'. In concordance with this, plans have arisen to exponentially scale up access to surgical care in low- and middle-income countries (LMICs). Children's surgery has yet to be formally recognised within these plans despite children forming up to 50% of the population in LMICs.

SSA has the highest unmet need for surgical care in the world at 41 million cases per year (29% of the worlds unmet need). 9% of the global surgical burden of disease is attributable to congenital anomalies. It is estimated that 2.6 million children are born with a congenital anomaly in SSA each year.

Hence, in order for the world to achieve the LCoGS goal of 80% coverage of surgical care by 2030, there must be a focus on scaling up neonatal and PS care in SSA where a significant proportion of the burden of surgical disease lies.

To date there has been limited data published on neonatal and PS in SSA. Nwomeh et al undertook a systematic review and meta-analysis of neonatal surgery in SSA and identified just 13 prospective studies and 38 retrospective studies between 1995 - 2014. The majority of these were single institutional studies, many with limited numbers. The results highlight poor outcomes with mortality rates of over 50-100% for conditions such as gastroschisis, which has mortality rates consistently under 4% in high-income countries. Similarly, the limited literature on PS in SSA highlights significantly poorer outcomes for common conditions such as appendicitis, intussusception and inguinal hernia.

Surgery has largely been overlooked in global health prioritisation and funding, likely because of the perception of prohibitive cost and complexity of care. Conversely, recent health economic studies have amply demonstrated the overall cost-effectiveness of PS procedures; for instance investing in a paediatric inguinal hernia repair is similar to administering a tetanus vaccine or treating a patient with malaria in terms of disability-adjusted life years (DALYS)/ US$.

This study aims to collect prospective data on five common neonatal and PS conditions across SSA, all of which have low morbidity and mortality (M&M) in high income countries (HICs), but reported poorer outcomes in SSA. It will be the first neonatal and PS cohort study across SSA and will undoubtedly form one of the largest prospective data sets in this region of the world.

The five conditions to be studied are gastroschisis, anorectal malformation, appendicitis, inguinal hernia and intussusception.

Gastroschisis

The incidence of gastroschisis is increasing worldwide, as are the number of these patients presenting to hospital in SSA. In Pretoria, South Africa, there was a 35-fold increase in patients presenting with gastroschisis from the early 1980's to late 1990s. Centres such as Harare, Zimbabwe, report receiving up to 3-4 cases per week. The true incidence of gastroschisis is unknown in SSA, however studies suggest the incidence, at least in some regions, appears to be similar to HICs. With a prevalence of 5.4/10,000 births, we can estimate that 1440 cases will be born each month in SSA.

Mortality rates for gastroschisis have fallen dramatically in HICs from 60% in the 1960's to less than 4% today. This has resulted from improvements in neonatal resuscitation and peri-operative management, awareness of complications such as abdominal compartment syndrome, and the provision of parenteral nutrition (PN). Gastroschisis has been suggested as a bellwether procedure for neonatal surgery capacity in low resource settings because there are usually no co-morbidities, yet the condition tests all the key elements that go into the successful management of a newborn with a surgical condition.

The data available regarding gastroschisis in SSA suggests significantly poorer outcomes than in HIC. Mortality rates have been reported as: 60% Malawi, 57-75% Nigeria, 84-100% Zimbabwe, 100% Uganda, 100% Cote'd'Ivoire. Mortality in South Africa is lower at 12-43%. In an international survey of gastroschisis, two thirds of the 25 institutions in SSA stated their mortality rate was >75% and the remaining third stated it was between 50-75%.

There is great variation in the management of gastroschisis across the globe and even between surgeons within the same institution. Primary closure rates vary from 16%, particularly in centres where routine use of preformed silos (PFS) have been adopted, to 92%. The majority of staged closure in SSA is undertaken using a surgical silo; PFS are utilised less due to lack of availability and training. Some surgeons recommend primary palliative care in SSA. A randomised control trial of primary closure versus PFS has reported they have similar outcomes, however there is a trend towards fewer ventilator days with the latter. A meta-analysis highlighted that the studies with least selection bias show that PFS is associated with fewer ventilator days (P<0.0001), reduced time to first feed (p=0.04) and lower infection rates (p=0.03).

There are many challenges faced by a surgeon in SSA. Patients are often outborn with no antenatal diagnosis, and hence presentation is delayed resulting in hypothermia, sepsis, hypovolaemia and bowel compromise. There is a natural tendency for babies with gastroschisis to be born early; in Harare 43% were preterm and 72% were <2.5kg. Similarly in Durban 64% were preterm and 72% <2.5kg. Many centres lack a neonatal intensive care unit (NICU) and have limited anaesthetic resources. Exposure of the bowel to amniotic fluid results in dysmotility and problems with absorption of nutrients; in the UK the average duration of parenteral (PN) requirement in simple gastroschisis is 23 days and 51 days in complex gastroschisis (gastroschisis associated with bowel perforation, necrosis or atresia). PN was only available in 36% of SSA centres when surveyed. However, in Harare the median hospital stay was 4.5days for the 85% who died, suggesting death was related to inadequate resuscitation and support rather than lack of PN. A multi-centre Gastroschisis International (GiT) study showed septicaemia to be the leading cause of death.

Some centres such as the University of Nigeria Teaching Hospital have introduced a protocol to ensure efficient pre- and post-operative resuscitation and care, preservation of body heat, decompression of the stomach with a nasogastric tube, evacuation of meconium, respiratory support and parental nutrition. As a result their mortality rate has fallen from 65% to 35%. However, Hadley notes that in Durban, despite access to NICU and PN, the overall mortality is still 43%, with sepsis being the leading cause of death. They stress the importance of meticulous central line care and a need for improved antenatal care and delivery within a tertiary paediatric surgery centre. A protocol focussed on early and aggressive resuscitation, avoidance of compartment syndrome, appropriate IV access and proactive nutritional interventions may help SSA start to realise the improvements in outcome as seen in HIC over the last 55-years. Implementing such interventions should have a knock on effect to strengthen the neonatal healthcare system in SSA and hence help to improve outcomes for all newborns with surgical conditions.

Anorectal Malformation

The birth prevalence of anorectal malformations (ARMs) has been reported as 1:1,500 - 1:5,000 in South Africa. In institutional publications from around SSA, caseload varies from 1-3 cases/ month. ARMs are one of the most common neonatal emergencies presenting to hospitals in SSA: 9.5% surgical neonates in Tanzania, 13.4% congenital malformations in Nigeria.

Mortality in HIC has fallen from 23% in the 1940's to less than 3% today. Mortality has been documented at 18.5 - 20% in Nigeria, with most deaths related to overwhelming sepsis, respiratory insufficiency and cyanotic heart disease. Unlike gastroschisis, 50% cases are associated with other anomalies: VACTERL (vertebral, anorectal, cardiac, tracheoesophageal, renal and limb). Other challenges include late presentation (2-5 days), low birth weight (38% < 2.5kg) and lack of adequate NICU facilities.

Management is dependent on the type of anomaly with low ARM typically being managed with a primary anoplasty and higher anomalies requiring a primary colostomy followed by a posterior sagittal anorectoplasty (PSARP) within the first year of life, and subsequent colostomy closure. Divided sigmoid colostomy is preferred to avoid overspill of stool from the proximal limb into the distal pouch, however some centres in SSA undertake loop colostomies. Lukong et al highlighted their improvement in outcome following a change in practice from a transverse loop colostomy to divided sigmoid colostomy with delayed PSARP. In some centres local anaesthesia is utilised to undertake the colostomy, reducing the risks associated with general anaesthesia where resources are limited.

Udefiagbon et al, highlight the problems with a colostomy, particularly in a low income setting: skin excoriation, wound infection, sepsis, prolapse, fluid and electrolyte losses and poor acceptance by care givers. They present impressive outcomes for primary PSARP undertaken during the first week of life. Authors advocate the benefits of reduced infection rate due to the sterile nature of the meconium and avoidance of a prolonged 3-stage procedure, which is more expensive and often unfeasible for African families. However, this practice requires safe neonatal anaesthesia, skilled surgeons and good standards of peri-operative care. Olivieri et al have described a modified PSARP technique utilised in Eritrea to reduce the risk of perianal wound infection where they leave a 3cm rectal stump, which is trimmed after 2 weeks. Poenaru et al advocate performing a wider anoplasty, which is less prone to stenosis, as regular dilatation and following-up can be challenging in this context.

This study will capture the primary peri-operative management and outcomes for patients presenting with ARM. Longer-term morbidity including faecal incontinence, anal stenosis, constipation, urinary and ejaculatory problems and outcomes of subsequent surgery are beyond the remit of this study.

Appendicitis

Acute appendicitis is one of the commonest causes for acute abdomen in children worldwide. In Ethiopia appendicitis accounts for 12% of emergency paediatric surgery and in the Congo it constitutes 30% of paediatric visceral surgery. Mortality from appendicitis is up to 4% in some SSA settings and morbidity high with wound infection rates up to 60% and wound dehiscence in up to 25%. Conversely, mortality from appendicitis in HICs is 0.04% and only 0.006% in children aged 9-19years. The LCoGS has listed laparotomy as one of three bellwether procedures that must be safe and available at all institutions providing first level care.

There are a number of challenges for managing children with acute appendicitis in the SSA setting. Children present late with 25-67% perforation rates; re-operation for intra-abdominal sepsis is as high as 40%. Differential diagnoses in SSA are more varied. In America, 82% of peritonitis in children is secondary to appendicitis whereas in SSA children present with peritonitis secondary to typhoid perforation, tuberculosis and ascariasis. There is often a lack of appropriate antibiotics, paediatric intensive care, blood products and parental nutrition. HIV may impact on the spectrum and severity of surgical infection in African children.

Inguinal Hernia

Paediatric inguinal hernia repair (PIHR) is the most commonly performed operation worldwide. The incidence is up to 5% of term infants and 30% of preterm. It is widely considered a basic and essential procedure that should be available to all and yet is largely unavailable in SSA. Complicated inguinal hernias pose a threat to the life of the child and considerable morbidity, which could be avoided by timely management of what is otherwise a straightforward procedure. Infants are at greatest risk of delay; Zamakhshary found that waiting over 2 weeks for a PIHR doubled the risk of incarceration in this age group.

In Ein's study of 6361 paediatric inguinal hernia repairs in Canada there were no deaths, recurrence rate of 1.2%, wound infection rate of 1.2% and testicular atrophy rate of 0.3%. In this study, 12% presented as incarcerated, but only 1% required emergency surgery for an irreducible hernia and 2/6361 required a bowel resection. Ergogan reported similar outcomes in Turkey.

In SSA, delays in presentation and lack of surgical capacity often result in a higher proportion of complicated paediatric hernias. In Nigeria, outcomes have been reported as: mortality 2.4%, intestinal resection 7%, testicular gangrene 15% and wound infection 15%. Another centre reported that in their cohort of infants presenting <42days of age, 52% were incarcerated, 36% required a bowel resection and 18% underwent an orchidectomy for testicular infarction. Strangulated hernias constitute 22% of the emergency visceral surgery in the Democratic Republic of the Congo. A randomised controlled trial in Nigeria reported a reduction in infection rate following PIHR from 4.8% to 0% with the use of prophylactic IV gentamycin at induction.

Intussusception

Intussusception is a leading cause of intestinal obstruction (IO) in children. A study from Nigeria reported 29% of IO from intussusception, 22% from ARM and 17% from obstructed PIH. The incidence is South Africa is comparable to HICs at 56/100,000 < 1-year compared to 33-49/100,000 < 1-year in the US. Published studies suggest institutions in SSA see at least one case/ month.

In HIC mortality is low at 0.1% in Europe and 0.4% in the US. Mortality rates in SSA vary widely and have been reported at 0 - 55%. The average mortality rate across SSA is 9.4%. There are a number of challenges to managing a child with intussusception in SSA. They often present late; 92% patients in Ile-Ife, Nigeria, present >24 hours. In Kenya the main duration of symptoms at presentation was 5 days (1-14). It was noted that the median delay for those who died (6.4%) was 5-days versus 3-days in those who survived. Surgical site infections following laparotomy for intussusception have been reported as high as 37.5%.

Management varies widely in SSA. In HICs most centres undertake air enema reduction (AER) as primary management in cases without peritonitis, perforation or non-responsive shock. This has been shown to be 1.48 times more effective than hydrostatic reduction (61% and 44% respectively). Centres in SSA with access to AER report good success rates; in a study in Ghana AER was successful in 59-67% cases and their mortality rate was 2%. They note that AER costs 20% of the fee for surgical management. A study from Nigeria reports offering hydrostatic reduction to 40% of cases, where it is successful in 64%. They also highlight the significant cost savings.

Ahmed et al in Egypt describe their simple AER equipment with a pressure release value at 120mmHg. They report an 88.2% success rate with no complications. Wiersma and Hadley advocate the use of AER in the operating theatre, which has improved their reduction rate to 53% from 22%.

Aim:

To compare outcomes of five common neonatal and paediatric surgical conditions between SSA and HICs.

Objectives:

1. To undertake the first multi-centre prospective cohort study across SSA to compare outcomes of common paediatric surgical conditions with benchmark data from HICs.
2. To identify context appropriate interventions and peri-operative factors associated with an improved outcome.
3. To form a research collaboration of paediatric surgeons and allied health professionals across SSA and help to enhance research capacity.
4. To raise awareness and provide advocacy for neonatal and paediatric surgical care within global health prioritisation, planning and funding.

Methodology

Authorship:

PaedSurg Africa constitutes a network of surgeons and allied health professionals who work with children requiring surgery across sub-Saharan Africa. This methodology is based on an equal partnership model previously described in the Lancet and utilised by a number of national and international collaboratives.

Publishing journals will be asked to make all co-authors PubMed citable. Articles will be published under 'PaedSurg Africa Research Collaboration'. At the end of the article co-authors will be listed under the following headings:

* Lead investigators: collaborators who have contributed to the study protocol, data analysis and write-up of the manuscript.
* Country leads: collaborators who have recruited several sites in their country to contribute to the study.
* Local investigators: collaborators who have gained ethical approval for the protocol in their centre and collected data at their site including patient identification and data completion with follow-up of mortality and complications.

The study invites up to three local investigators per institution per month of data collection.

Collaborator Recruitment:

Primary recruitment will be through the lead investigators' personal contacts, which span many centres and countries across SSA, and the Pan-African Paediatric Surgical Association (PAPSA) mailing list. Research collaborators were recruited at the Global Initiative for Children's Surgery (GICS) Conference hosted by the Royal College of Surgeons of England, May 2016. A further recruitment drive will be undertaken at the PAPSA Conference in Nigeria (September 2016) where the research proposal will be presented, investigators actively sought, and REDCap sign-up, app download and project set-up achieved.

Data Collection Tool:

Prospective data will be collected over a 1-month period utilising the free, user-friendly, secure database, REDCap. The tool includes a Smartphone app that allows offline data collection. Data collection sheets that can be printed for written data collection and later uploaded will also be provided. Data collection will be open for any continuous 1-month period between October 2016 to April 2017, to optimise uptake. A pilot study will be run in August/ September 2016 at five institutions in SSA.

Conditions Studied:

The five conditions selected are common congenital or acquired neonatal and paediatric surgical conditions with low morbidity and mortality in HICs. Consequently surgical interventions for these conditions carry high avertable DALYs and cost-effectiveness ratios, as saving the life of a neonate or child with minimal long-term disability can permit a lifetime of labour and income for their family and their country's economy. Limited, mostly retrospective, individual institutional studies suggest significantly poorer outcomes of these conditions in SSA.

Validation:

At 5% of collaborating centres, one additional research collaborator will be asked to identify patients and upload the study data independent to the other research collaborator(s) at their centre. This data will be collected on a separate REDCap validation database and the inputted data will be cross-checked with that entered into the main database. Only patients with over 90% of data inputted will be included in the study. Data can be initially uploaded and completed at a later date prior to submission if any data is missing.

Questionnaire Data:

A short questionnaire will be undertaken by all research collaborators at the time of project sign up regarding the facilities and resources available at their institution.

Estimated Population:

Estimated patient numbers per centre during a 1-month study period are: 1-2 gastroschisis, 1-2 anorectal malformations, 11 appendicitis, 14 inguinal hernias, 1 intussusception (29 patients per centre). We aim to include a minimum of 50 centres, which would generate 1450 patients. Estimates were calculated using the mean number of patients presenting per month to all institutions from SSA who have published data on these conditions.

Data Analysis:

Power calculations were undertaken to determine the minimum detectable differences in mortality between SSA and benchmark data from HICs. These confirm that the study is adequately powered to detect a difference in mortality of each of the five conditions between SSA and HICs at a 5% significance level and 80% power. Outcomes in SSA compared to HICs will be presented as relative risks and significant differences determined using Chi-Squared analysis.

Multi-level, multivariate logistic regression analysis will be utilised to identify context appropriate interventions and peri-operative factors associated with improved outcomes. For example: does availability of air enema reduction significantly reduce mortality from intussusception in the SSA context and if so, by how much? Results will be presented as odds ratios. Data will be adjusted for confounding factors such as delay in presentation. P<0.05 will be deemed significant.

Ethics:

Full ethical approval for the project has been granted by the host centre, Kings College London Research Ethics Committee. Research collaborators in SSA will be required to receive approval for the project at their own centres according to local ethical regulations and provide evidence of this in order to submit data.

If no formal ethics or audit committee exists, collaborators must provide written consent from the Director of the Hospital or Head of Surgical Department. All data will be anonymous. Data will not be identifiable at individual surgeon, institution or country level.

Outcome:

The results from this study can be used to advocate for enhanced neonatal and paediatric surgical care in SSA, at an institutional level, country level via 'National Health Strategic Plans' and at an international level. This is vital to ensure neonatal and paediatric surgery are appropriately prioritised over the coming 15-years as access to surgical care in low- and middle-income countries is scaled up following publication of the LCoGS and the WHA resolution 68:15. Participation in this international project will help to enhance research capacity amongst surgeons, anaesthetists and allied healthcare professionals across SSA. Formation of the PaedSurg Africa Research Collaboration will provide the infrastructure for future research projects and interventional studies to help improve outcome.

ELIGIBILITY:
Inclusion Criteria:

All patients under 16-years of age presenting primarily with one of the five study conditions during the data collection period. This includes those managed conservatively without surgery or intervention and those offered palliative care, except patients with an inguinal hernia who must receive surgery to be included.

Exclusion Criteria:

Patients re-presenting with one of the five study conditions with a complication from a previous intervention or requiring further surgical intervention.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Collaborating centres were recruited using convenience sampling with snowballing. Centres include both tertiary paediatric surgery centres and district hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1407 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
All-cause in-hospital mortality | In-hospital (if in the patient is still in hospital at 30-days post-intervention, a 30-day mortality will be utilised)

SECONDARY OUTCOMES:
30-day mortality | 30-days
  Whether or not the patient died within 30-days of intervention
Duration of hospital stay | Patients are followed up for a maximum of 30-days post-intervention
  Total number of days in hospital inclusive of the day of admission and day of discharge
Surgical site infection | Within 30-days post-intervention
  Surgical site infection criteria include at least one of the following: 1) purulent drainage from the superficial or deep (fascia or muscle) incision but not from within the organ/space component of the surgical site, 2) at least one of: pain or tenderness; localised swelling; redness; heat; fever; AND the incision is opened deliberately or spontaneously dehisces, 3) there is an abscess within the wound (clinically or radiologically detected).
Full thickness wound dehiscence | Within 30-days post-intervention
  This is defined as all wound layers opening.
Need for re-intervention | Within 30-days of the primary intervention
  Including surgical or percutaneous intervention

CONTACTS AND LOCATIONS:
Locations (1):
- King's Centre for Global Health and Health Partnerships, Denmark Hill, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following publication, the full anonymous data set will be made publicly available.

REFERENCES:
- [Background] GlobalSurg Collaborative. Mortality of emergency abdominal surgery in high-, middle- and low-income countries. Br J Surg. 2016 Jul;103(8):971-988. doi: 10.1002/bjs.10151. Epub 2016 May 4. PMID 27145169
- [Background] Poenaru D, Pemberton J, Frankfurter C, Cameron BH. Quantifying the Disability from Congenital Anomalies Averted Through Pediatric Surgery: A Cross-Sectional Comparison of a Pediatric Surgical Unit in Kenya and Canada. World J Surg. 2015 Sep;39(9):2198-206. doi: 10.1007/s00268-015-3103-8. PMID 26037026
- [Background] Price R, Makasa E, Hollands M. World Health Assembly Resolution WHA68.15: "Strengthening Emergency and Essential Surgical Care and Anesthesia as a Component of Universal Health Coverage"-Addressing the Public Health Gaps Arising from Lack of Safe, Affordable and Accessible Surgical and Anesthetic Services. World J Surg. 2015 Sep;39(9):2115-25. doi: 10.1007/s00268-015-3153-y. PMID 26239773
- [Background] Ekenze SO, Ajuzieogu OV, Nwomeh BC. Challenges of management and outcome of neonatal surgery in Africa: a systematic review. Pediatr Surg Int. 2016 Mar;32(3):291-9. doi: 10.1007/s00383-016-3861-x. Epub 2016 Jan 18. PMID 26783085
- [Background] Bradnock TJ, Marven S, Owen A, Johnson P, Kurinczuk JJ, Spark P, Draper ES, Knight M; BAPS-CASS. Gastroschisis: one year outcomes from national cohort study. BMJ. 2011 Nov 15;343:d6749. doi: 10.1136/bmj.d6749. PMID 22089731
- [Background] Ademola TO, Oludayo SA, Samuel OA, Amarachukwu EC, Akinwunmi KO, Olusanya A. Clinicopathological review of 156 appendicectomies for acute appendicitis in children in Ile-Ife, Nigeria: a retrospective analysis. BMC Emerg Med. 2015 May 9;15:7. doi: 10.1186/s12873-015-0030-9. PMID 25956068
- [Background] Hadley GP. Intra-abdominal sepsis--epidemiology, aetiology and management. Semin Pediatr Surg. 2014 Dec;23(6):357-62. doi: 10.1053/j.sempedsurg.2014.06.008. Epub 2014 Jun 4. PMID 25459442
- [Background] Ameh EA, Abantanga FA, Birabwa-Male D. Surgical aspects of bacterial infection in African children. Semin Pediatr Surg. 2012 May;21(2):116-24. doi: 10.1053/j.sempedsurg.2012.01.004. PMID 22475117
- [Background] Bamigbola KT, Nasir AA, Abdur-Rahman LO, Adeniran JO. Complicated childhood inguinal hernias in UITH, Ilorin. Afr J Paediatr Surg. 2012 Sep-Dec;9(3):227-30. doi: 10.4103/0189-6725.104725. PMID 23250245
- [Background] Mabiala-Babela JR, Pandzou N, Koutaba E, Ganga-Zandzou S, Senga P. [Retrospective study of visceral surgical emergencies in children at the University Hospital Center of Brazzaville (Congo)]. Med Trop (Mars). 2006 Apr;66(2):172-6. French. PMID 16775942
- [Background] Jiang J, Jiang B, Parashar U, Nguyen T, Bines J, Patel MM. Childhood intussusception: a literature review. PLoS One. 2013 Jul 22;8(7):e68482. doi: 10.1371/journal.pone.0068482. Print 2013. PMID 23894308
- [Background] Eeson G, Birabwa-Male D, Pennington M, Blair GK. Costs and cost-effectiveness of pediatric inguinal hernia repair in Uganda. World J Surg. 2015 Feb;39(2):343-9. doi: 10.1007/s00268-014-2818-2. PMID 25270348
- [Background] Citron I, Chokotho L, Lavy C. Prioritisation of surgery in the National Health Strategic Plans of Africa: a systematic review. Lancet. 2015 Apr 27;385 Suppl 2:S53. doi: 10.1016/S0140-6736(15)60848-0. Epub 2015 Apr 26. PMID 26313103
- [Background] Agugua NE, Nwako FA. Gastroschisis a fifteen-year experience. West Afr J Med. 1990 Apr-Jun;9(2):147-50. PMID 2148495
- [Background] Arnold M. Is the incidence of gastroschisis rising in South Africa in accordance with international trends? A retrospective analysis at Pretoria Academic and Kalafong Hospitals, 1981-2001. S Afr J Surg. 2004 Aug;42(3):86-8. PMID 15532615
- [Background] Wright NJ, Zani A, Ade-Ajayi N. Epidemiology, management and outcome of gastroschisis in Sub-Saharan Africa: Results of an international survey. Afr J Paediatr Surg. 2015 Jan-Mar;12(1):1-6. doi: 10.4103/0189-6725.150924. PMID 25659541
- [Background] Ford K, Poenaru D, Moulot O, Tavener K, Bradley S, Bankole R, Tshifularo N, Ameh E, Alema N, Borgstein E, Hickey A, Ade-Ajayi N. Gastroschisis: Bellwether for neonatal surgery capacity in low resource settings? J Pediatr Surg. 2016 Aug;51(8):1262-7. doi: 10.1016/j.jpedsurg.2016.02.090. Epub 2016 Mar 12. PMID 27032610
- [Background] Iliff PJ. Neonatal surgery in Harare Hospital. Cent Afr J Med. 1990 Jan;36(1):11-5. PMID 2397493
- [Background] Apfeld JC, Wren SM, Macheka N, Mbuwayesango BA, Bruzoni M, Sylvester KG, Kastenberg ZJ. Infant, maternal, and geographic factors influencing gastroschisis related mortality in Zimbabwe. Surgery. 2015 Dec;158(6):1475-80. doi: 10.1016/j.surg.2015.04.037. Epub 2015 Jun 11. PMID 26071924
- [Background] Abdur-Rahman LO, Abdulrasheed NA, Adeniran JO. Challenges and outcomes of management of anterior abdominal wall defects in a Nigerian tertiary hospital. Afr J Paediatr Surg. 2011 May-Aug;8(2):159-63. doi: 10.4103/0189-6725.86053. PMID 22005356
- [Background] Sekabira J, Hadley GP. Gastroschisis: a third world perspective. Pediatr Surg Int. 2009 Apr;25(4):327-9. doi: 10.1007/s00383-009-2348-4. Epub 2009 Mar 14. PMID 19288118
- [Background] Davies MR, Beale PG. The pivotal role of the surgeon in the results achieved in gastroschisis. Pediatr Surg Int. 1996 Mar;11(2-3):82-5. doi: 10.1007/BF00183731. PMID 24057522
- [Background] Zani A, Ruttenstock E, Davenport M, Ade-Ajayi N. Is there unity in Europe? First survey of EUPSA delegates on the management of gastroschisis. Eur J Pediatr Surg. 2013 Feb;23(1):19-24. doi: 10.1055/s-0032-1326954. Epub 2012 Oct 23. PMID 23093440
- [Background] Weil BR, Leys CM, Rescorla FJ. The jury is still out: changes in gastroschisis management over the last decade are associated with both benefits and shortcomings. J Pediatr Surg. 2012 Jan;47(1):119-24. doi: 10.1016/j.jpedsurg.2011.10.029. PMID 22244403
- [Background] Pastor AC, Phillips JD, Fenton SJ, Meyers RL, Lamm AW, Raval MV, Lehman E, Karp TB, Wales PW, Langer JC. Routine use of a SILASTIC spring-loaded silo for infants with gastroschisis: a multicenter randomized controlled trial. J Pediatr Surg. 2008 Oct;43(10):1807-12. doi: 10.1016/j.jpedsurg.2008.04.003. PMID 18926212
- [Background] Kunz SN, Tieder JS, Whitlock K, Jackson JC, Avansino JR. Primary fascial closure versus staged closure with silo in patients with gastroschisis: a meta-analysis. J Pediatr Surg. 2013 Apr;48(4):845-57. doi: 10.1016/j.jpedsurg.2013.01.020. PMID 23583145
- [Background] Theron A, Loveland J. Birth prevalence of anorectal malformation in the referral area for the University of the Witwatersrand tertiary hospitals, South Africa. Eur J Pediatr Surg. 2015 Apr;25(2):220-5. doi: 10.1055/s-0033-1360456. Epub 2014 Feb 10. PMID 24515733
- [Background] Safavi A, Skarsgard E, Butterworth S. Bowel-defect disproportion in gastroschisis: does the need to extend the fascial defect predict outcome? Pediatr Surg Int. 2012 May;28(5):495-500. doi: 10.1007/s00383-012-3055-0. Epub 2012 Feb 14. PMID 22331201
- [Background] Govender S, Wiersma R. Delayed diagnosis of anorectal malformations (ARM): causes and consequences in a resource-constrained environment. Pediatr Surg Int. 2016 Apr;32(4):369-75. doi: 10.1007/s00383-016-3866-5. Epub 2016 Jan 20. PMID 26790675
- [Background] Kigo CN, Ndung'u JM. Bowel function following primary repair of anorectal malformations at Kenyatta National Hospital. East Afr Med J. 2002 Mar;79(3):124-7. doi: 10.4314/eamj.v79i3.8889. PMID 12389955
- [Background] Chirdan LB, Uba FA, Ameh EA, Mshelbwala PM. Colostomy for high anorectal malformation: an evaluation of morbidity and mortality in a developing country. Pediatr Surg Int. 2008 Apr;24(4):407-10. doi: 10.1007/s00383-008-2114-z. Epub 2008 Feb 13. PMID 18270719
- [Background] Lawal TA, Olulana DI, Ogundoyin OO. Spectrum of colorectal surgery operations performed in a single paediatric surgery unit in sub-Saharan Africa. Afr J Paediatr Surg. 2014 Apr-Jun;11(2):128-31. doi: 10.4103/0189-6725.132802. PMID 24841012
- [Background] Olivieri C, Belay K, Coletta R, Retrosi G, Molle P, Calisti A. Preventing posterior sagittal anoplasty 'cripples' in areas with limited medical resources: a few modifications to surgical approach in anorectal malformations. Afr J Paediatr Surg. 2012 Sep-Dec;9(3):223-6. doi: 10.4103/0189-6725.104724. PMID 23250244
- [Background] Nandi B, Mungongo C, Lakhoo K. A comparison of neonatal surgical admissions between two linked surgical departments in Africa and Europe. Pediatr Surg Int. 2008 Aug;24(8):939-42. doi: 10.1007/s00383-008-2177-x. Epub 2008 Jun 14. PMID 18553088
- [Background] Adeyemo AA, Gbadegesin RA, Omotade OO. Major congenital malformations among neonatal referrals to a Nigerian university hospital. East Afr Med J. 1997 Nov;74(11):699-701. PMID 9557439
- [Background] Ameh EA, Chirdan LB. Neonatal intestinal obstruction in Zaria, Nigeria. East Afr Med J. 2000 Sep;77(9):510-3. doi: 10.4314/eamj.v77i9.46702. PMID 12862145
- [Background] Shah M, Gallaher J, Msiska N, McLean SE, Charles AG. Pediatric intestinal obstruction in Malawi: characteristics and outcomes. Am J Surg. 2016 Apr;211(4):722-6. doi: 10.1016/j.amjsurg.2015.11.024. Epub 2016 Jan 6. PMID 26810940
- [Background] Rintala RJ, Pakarinen MP. Imperforate anus: long- and short-term outcome. Semin Pediatr Surg. 2008 May;17(2):79-89. doi: 10.1053/j.sempedsurg.2008.02.003. PMID 18395657
- [Background] Lukong CS, Ameh EA, Mshelbwala PM, Jabo BA, Gomna A, Akiniyi OT, Nmadu PT. Management of anorectal malformation: Changing trend over two decades in Zaria, Nigeria. Afr J Paediatr Surg. 2011 Jan-Apr;8(1):19-22. doi: 10.4103/0189-6725.78663. PMID 21478581
- [Background] Osifo OD, Osagie TO, Udefiagbon EO. Outcome of primary posterior sagittal anorectoplasty of high anorectal malformation in well selected neonates. Niger J Clin Pract. 2014 Jan-Feb;17(1):1-5. doi: 10.4103/1119-3077.122821. PMID 24326797
- [Background] Poenaru D, Borgstein E, Numanoglu A, Azzie G. Caring for children with colorectal disease in the context of limited resources. Semin Pediatr Surg. 2010 May;19(2):118-27. doi: 10.1053/j.sempedsurg.2009.11.017. PMID 20307848
- [Background] Derbew M, Ahmed E. The pattern of pediatric surgical conditions in Tikur Anbessa Unversity Hospital, Addis Ababa, Ethiopia. Ethiop Med J. 2006 Oct;44(4):331-8. PMID 17370432
- [Background] Momoh JT. External hernia in Nigerian children. Ann Trop Paediatr. 1985 Dec;5(4):197-200. doi: 10.1080/02724936.1985.11748392. PMID 2418768
- [Background] Daniel E, Mersha D. Childhood appendicitis: factors associated with its incidence and perforation in Ethiopian children. Ethiop Med J. 1991 Jan;29(1):15-9. PMID 2001686
- [Background] Ein SH, Njere I, Ein A. Six thousand three hundred sixty-one pediatric inguinal hernias: a 35-year review. J Pediatr Surg. 2006 May;41(5):980-6. doi: 10.1016/j.jpedsurg.2006.01.020. PMID 16677897
- [Background] Ohene-Yeboah M, Abantanga FA. Inguinal hernia disease in Africa: a common but neglected surgical condition. West Afr J Med. 2011 Mar-Apr;30(2):77-83. PMID 21984452
- [Background] Zamakhshary M, To T, Guan J, Langer JC. Risk of incarceration of inguinal hernia among infants and young children awaiting elective surgery. CMAJ. 2008 Nov 4;179(10):1001-5. doi: 10.1503/cmaj.070923. PMID 18981440
- [Background] Erdogan D, Karaman I, Aslan MK, Karaman A, Cavusoglu YH. Analysis of 3,776 pediatric inguinal hernia and hydrocele cases in a tertiary center. J Pediatr Surg. 2013 Aug;48(8):1767-72. doi: 10.1016/j.jpedsurg.2012.09.048. PMID 23932620
- [Background] Ameh EA. Morbidity and mortality of inguinal hernia in the newborn. Niger Postgrad Med J. 2002 Dec;9(4):233-4. PMID 12690685
- [Background] Usang UE, Sowande OA, Adejuyigbe O, Bakare TI, Ademuyiwa OA. The role of preoperative antibiotics in the prevention of wound infection after day case surgery for inguinal hernia in children in Ile Ife, Nigeria. Pediatr Surg Int. 2008 Oct;24(10):1181-5. doi: 10.1007/s00383-008-2241-6. Epub 2008 Aug 23. PMID 18726104
- [Background] Ogundoyin OO, Afolabi AO, Ogunlana DI, Lawal TA, Yifieyeh AC. Pattern and outcome of childhood intestinal obstruction at a tertiary hospital in Nigeria. Afr Health Sci. 2009 Sep;9(3):170-3. PMID 20589146
- [Background] Stolz LA, Kizza H, Little K, Kasekende J. Intussusception detected with ultrasound in a resource-limited setting. Lancet. 2013 Jun 8;381(9882):2054. doi: 10.1016/S0140-6736(13)60690-X. No abstract available. PMID 23746905
- [Background] Omore R, Osawa F, Musia J, Rha B, Ismail A, Kiulia NM, Moke F, Vulule J, Wainaina AM, Tole J, Machoki SM, Nuorti JP, Breiman RF, Parashar UD, Montgomery JM, Tate JE. Intussusception Cases Among Children Admitted to Referral Hospitals in Kenya, 2002-2013: Implications for Monitoring Postlicensure Safety of Rotavirus Vaccines in Africa. J Pediatric Infect Dis Soc. 2016 Dec;5(4):465-469. doi: 10.1093/jpids/piv051. Epub 2015 Aug 25. PMID 26407281
- [Background] Talabi AO, Sowande OA, Etonyeaku CA, Adejuyigbe O. Childhood intussusception in Ile-ife: what has changed? Afr J Paediatr Surg. 2013 Jul-Sep;10(3):239-42. doi: 10.4103/0189-6725.120900. PMID 24192467
- [Background] Mpabalwani EM, Chitambala P, Chibumbya JN, Matapo B, Mutambo H, Mwenda JM, Babaniyi O, Munkonge L. Intussusception incidence rates in 9 Zambian hospitals, 2007-2011: prerotavirus vaccine introduction. Pediatr Infect Dis J. 2014 Jan;33 Suppl 1:S94-8. doi: 10.1097/INF.0000000000000055. PMID 24343623
- [Background] Steele AD, Patel M, Cunliffe NA, Bresee JS, Borgstein E, Parashar UD. Workshop on intussusception in African countries--meeting report. Vaccine. 2012 Apr 27;30 Suppl 1:A185-9. doi: 10.1016/j.vaccine.2011.10.004. PMID 22520130
- [Background] Moore SW, Kirsten M, Muller EW, Numanoglu A, Chitnis M, Le Grange E, Banieghbal B, Hadley GP. Retrospective surveillance of intussusception in South Africa, 1998-2003. J Infect Dis. 2010 Sep 1;202 Suppl:S156-61. doi: 10.1086/653563. PMID 20684696
- [Background] Abantanga FA, Amoah M, Adeyinka AO, Nimako B, Yankey KP. Pneumatic reduction of intussusception in children at the Komfo Anokye Hospital, Kumasi, Ghana. East Afr Med J. 2008 Nov;85(11):550-5. doi: 10.4314/eamj.v85i11.9672. PMID 19413208
- [Background] Kuremu RT. Childhood intussusception at the Moi teaching and Referral Hospital Eldoret: management challenges in a rural setting. East Afr Med J. 2004 Sep;81(9):443-6. doi: 10.4314/eamj.v81i9.9218. PMID 15626052
- [Background] Carneiro PM, Kisusi DM. Intussusception in children seen at Muhimbili National Hospital, Dar es Salaam. East Afr Med J. 2004 Sep;81(9):439-42. doi: 10.4314/eamj.v81i9.9217. PMID 15626051
- [Background] Edino ST, Ochicha O, Mohammed AZ, Anumah M. Intussusception in Kano: a 5-year analysis of pattern, morbidity and mortality. Niger J Med. 2003 Oct-Dec;12(4):221-4. PMID 14768198
- [Background] Ameh EA. The morbidity and mortality of right hemicolectomy for complicated intussusception in infants. Niger Postgrad Med J. 2002 Sep;9(3):123-4. PMID 12501272
- [Background] Ameh EA. The morbidity and mortality of laparotomy for uncomplicated intussusception in children. West Afr J Med. 2002 Apr-Jun;21(2):115-6. PMID 12403031
- [Background] Harouna Y, Tardivel G, Abdou I, Gamatie Y, Mariama S, Bia M. [Prognosis of acute intestinal intussusception in infants at the national hospital of Niamey (Niger). Eleven cases treated surgically]. Bull Soc Pathol Exot. 1997;90(1):30-2. French. PMID 9264747
- [Background] Adejuyigbe O, Jeje EA, Owa JA. Childhood intussusception in Ile-Ife, Nigeria. Ann Trop Paediatr. 1991;11(2):123-7. doi: 10.1080/02724936.1991.11747490. PMID 1715142
- [Background] Abdur-Rahman LO, Adeniran JO, Taiwo JO, Nasir AA, Odi T. Bowel resection in Nigerian children. Afr J Paediatr Surg. 2009 Jul-Dec;6(2):85-7. doi: 10.4103/0189-6725.54769. PMID 19661636
- [Background] Ogundoyin OO, Olulana DI, Lawal TA. Childhood intussusception: A prospective study of management trend in a developing country. Afr J Paediatr Surg. 2015 Oct-Dec;12(4):217-20. doi: 10.4103/0189-6725.172541. PMID 26712283
- [Background] Ekenze SO, Mgbor SO, Okwesili OR. Routine surgical intervention for childhood intussusception in a developing country. Ann Afr Med. 2010 Jan-Mar;9(1):27-30. doi: 10.4103/1596-3519.62621. PMID 20418646
- [Background] Carapinha C, Truter M, Bentley A, Welthagen A, Loveland J. Factors determining clinical outcomes in intussusception in the developing world: Experience from Johannesburg, South Africa. S Afr Med J. 2016 Jan 12;106(2):177-80. doi: 10.7196/SAMJ.2016.v106i2.9672. PMID 26821898
- [Background] Chalya PL, Kayange NM, Chandika AB. Childhood intussusceptions at a tertiary care hospital in northwestern Tanzania: a diagnostic and therapeutic challenge in resource-limited setting. Ital J Pediatr. 2014 Mar 11;40(1):28. doi: 10.1186/1824-7288-40-28. PMID 24618338
- [Background] Khorana J, Singhavejsakul J, Ukarapol N, Laohapensang M, Wakhanrittee J, Patumanond J. Enema reduction of intussusception: the success rate of hydrostatic and pneumatic reduction. Ther Clin Risk Manag. 2015 Dec 15;11:1837-42. doi: 10.2147/TCRM.S92169. eCollection 2015. PMID 26719697
- [Background] Mensah YB, Glover-Addy H, Etwire V, Twum MB, Asiamah S, Appeadu-Mensah W, Hesse AA. Pneumatic reduction of intussusception in children at Korle Bu Teaching Hospital: an initial experience. Afr J Paediatr Surg. 2011 May-Aug;8(2):176-81. doi: 10.4103/0189-6725.86057. PMID 22005360
- [Background] Ahmed HM, Ahmed O, Ahmed RK. Adding a custom made pressure release valve during air enema for intussusception: A new technique. Afr J Paediatr Surg. 2015 Oct-Dec;12(4):232-5. doi: 10.4103/0189-6725.172550. PMID 26712286
- [Background] Wiersma R, Hadley GP. Minimizing surgery in complicated intussusceptions in the Third World. Pediatr Surg Int. 2004 Mar;20(3):215-7. doi: 10.1007/s00383-003-1099-x. Epub 2004 Apr 3. PMID 15064960
- [Background] Bhangu A, Kolias AG, Pinkney T, Hall NJ, Fitzgerald JE. Surgical research collaboratives in the UK. Lancet. 2013 Sep 28;382(9898):1091-2. doi: 10.1016/S0140-6736(13)62013-9. No abstract available. PMID 24075040
- [Background] Kong VY, Sartorius B, Clarke DL. Acute appendicitis in the developing world is a morbid disease. Ann R Coll Surg Engl. 2015 Jul;97(5):390-5. doi: 10.1308/003588415X14181254790608. PMID 26264094
- [Background] Ameh EA. Incarcerated and strangulated inguinal hernias in children in Zaria, Nigeria. East Afr Med J. 1999 Sep;76(9):499-501. PMID 10685318
- [Background] Ohene-Yeboah M, Abantanga F, Oppong J, Togbe B, Nimako B, Amoah M, Azorliade R. Some aspects of the epidemiology of external hernias in Kumasi, Ghana. Hernia. 2009 Oct;13(5):529-32. doi: 10.1007/s10029-009-0491-4. Epub 2009 Mar 20. PMID 19301084
- [Background] Healy DA, Doyle D, Moynagh E, Maguire M, Ahmed I, Ahmed AS, Caldwell M, O'Hanrahan T, Walsh SR. Systematic Review and Meta-Analysis on the Influence of Surgeon Specialization on Outcomes Following Appendicectomy in Children. Medicine (Baltimore). 2015 Aug;94(32):e1352. doi: 10.1097/MD.0000000000001352. PMID 26266388
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686